CLINICAL TRIAL: NCT03089658
Title: Temporary Authorization for Use (ATU) to Avelumab for Treatment of Adult Patients With Metastatic Merkel Cell Carcinoma (mMCC)
Brief Title: Expanded Access to Avelumab for Treatment of Metastatic Merkel Cell Carcinoma (mMCC)
Status: Approved for marketing | Type: Expanded Access
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: MS100070_0308
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Metastatic Merkel Cell Carcinoma
Keywords: Metastatic Merkel Cell Carcinoma; Expanded Access Program; Temporary Authorisation for Use; Avelumab
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — avelumab

INTERVENTIONS:
Drug: Avelumab — Avelumab should be administered intravenously as per the recommended dose. Administration of Avelumab should continue according to the recommended schedule until disease progression or unacceptable toxicity.

SUMMARY:
Expanded access to Avelumab solution for infusion will be made available for adult patients with mMCC whose disease has progressed after receiving at least one prior chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Measurable metastatic Merkel cell carcinoma according to Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST v1.1), has failed at least one line of adequately dosed chemotherapy in the metastatic setting and has subsequently progressed (where adequate dosing is defined as a minimum of 2 cycles)
* Not eligible for participation in any ongoing clinical trial for Merkel cell carcinoma including the Javelin Merkel 200 study (NCT02155647)
* Adequate hematological, hepatic and renal function as defined in the protocol

Exclusion Criteria:

* Brain metastases
* Prior organ transplantation, including allogeneic stem cell transplantation
* History of testing positive for human immunodeficiency virus (HIV) or known AIDS or active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Concurrent, active, malignant disease (other than Merkel cell carcinoma) with the exception of basal or squamous cell carcinoma of the skin or carcinoma in situ as defined in protocol
* Previous or active autoimmune disease requiring systemic immunosuppressive therapy
* Known severe hypersensitivity reactions to monoclonal antibodies, any history of anaphylaxis, or uncontrolled asthma
* Clinically significant (that is, active) cardiovascular disease: cerebral vascular accident / stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment) unstable angina, congestive heart failure (New York Heart Association Classification Class ≥ II), or serious cardiac arrhythmia requiring medication
* Persisting toxicity related to prior therapy of Grade >1 NCI-CTCAE v 4.03 (alopecia and sensory neuropathy Grade ≤ 2 is acceptable)
* Being treated with chronic systemic corticosteroids or other chronic therapeutic immunosuppression
* Pregnant or lactating (for women of childbearing potential)
* Not using a highly effective contraception if the risk of conception exists

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Avelumab ATU Unit, Lyon, France